CLINICAL TRIAL: NCT04625582
Title: Modeling and Effectiveness of an Educational Intervention for the Development of Professional Skills in Family Medicine and Community Nurses Residents (PROEMPATIA)
Brief Title: Educational Intervention for the Development of Professionals Skills in Family Medicine and Community Nursing Residents
Acronym: PROEMPATHY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Galician South Health Research Institute (Network)
Collaborators: Aragon Health Science Institute (Other Government); Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: IISGS6/2020/11
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Empathy; Burnout, Professional
Keywords: Intervention study; Family Medicine trainees; Community Nursing trainees
MeSH Terms: conditions — Burnout, Professional | interventions — Pharmaceutical Services, Online

STUDY DESIGN:
Intervention Model Description: Ante-post evaluation study of the effectiveness of an educational intervention to improve empathy, with three arms: face-to-face, online and control group, lasting 2 years. The intervention is organized during the training of residents of Family Medicine and Community Nursing in three teaching units in different Spanish Health Authorities.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Face-to-face intervention (Experimental): 90 trainees at Vigo Family Medicine and Community Nursing Training Unit
  Interventions: Behavioral: Face-to-face
- Online intervention (Experimental): 70 trainees at Aragón Family Medicine and Community Nursing Training Unit
  Interventions: Behavioral: Online
- Usual training (No Intervention): 180 trainees at Balearic Islands Family Medicine and Community Nursing Training Unit

INTERVENTIONS:
Behavioral: Face-to-face — The intervention has been created specifically for this group of trainees, with the aim of acquiring or improving mediating personal skills in the processes of physical and mental well-being that help them cope with more motivation, enthusiasm and personal resources professional challenges.
  It is based on conducting 4-hour face-to-face workshops, every four months throughout the period of specialized health training. They will be instrumented through group dynamics, communication exercises, leadership, corporality, and reflective and emotional writing.
  Audiovisual media (videos, presentations, recordings) will be used. They will be developed in person in a classroom equipped with the necessary means for training, including versatility of the space.
  Arms: Face-to-face intervention
Behavioral: Online — The online intervention will pursue the same objectives and will be nourished by the same content as the face-to-face intervention. The theoretical content will be adapted for online use, with the flexibility of access and organization that this entails for the participants, including videos, presentations, recordings ...
  Group techniques will be carried out online, every four months during the entire period of specialized health professional training. They will be instrumented through group dynamics, communication exercises, leadership, corporality, and reflective and emotional writing.
  Arms: Online intervention

SUMMARY:
BACKGROUND The burnout syndrome among health care workers frequently rises to prevalence above 50%. One of the consequences most supported by the literature is the impoverishment of the therapeutic alliance, triggered by a loss of empathy of the clinician towards the patient due to the emotional exhaustion he or she suffers.

The main factors that influence the presence of this pathology are stressors related to the organization of work. However, this equation is also influenced by individual factors that can be acted upon and which are often the only tools available for professionals.

Due to the widely supported relationship of empathy, burnout and therapeutic alliance, the investigators decided to carry out a complex training plan focused on personal development in teaching units of Family and Community Care in Spain.

RESEARCH QUESTION Is effective an intervention aimed to promoting the development of personal skills throughout the training of family and community care doctors and nurses?

METHOD Pre-post study, comparing two educational interventions, one face-to-face (N=90) and other online (N=70), with a control group (N=170).

Participants: All physicians and nurse trainees on Primary Health Care in three Spanish Health Regions who wish to participate in the study. The face-to-face intervention consists of 3 annual workshops, while the online one will be carried out by adapting the theoretical contents of the face-to-face intervention for online use and will pursue the same objectives and be fed by the same contents.

The variation in the level of empathy will be quantified by means of the Interpersonal Reactivity Index (IRI) questionnaire, adjusted by burnout (Copenhagen questionnaire) and other variables such as resilience (Connor-Davidson), locus of control, social support (Oslo-3), sense of coherence (OLQ-13), age, sex, personality (Ten Item Personality Inventory, TIPI-SP) and other organisational factors.

Statistical analysis with generalized lineal models and generalized additive models.

DETAILED DESCRIPTION:
With the purpose of modeling and evaluating a comprehensive personal development intervention in family and community care residents (doctors and nurses) this project is proposed. With two expected results from the professionals' perspective: first, to evaluate the changes in self-perceived empathy; on the other hand, the modification of the level of exhaustion in them. In both, taking into account the personal factors discussed above, as well as organizational or training factors during this period of the residents' lives.

In essence, our model assumes that personal (on which the intervention will act) and organizational factors modulate changes in the exhaustion of residents during their residence. In turn, the differences in professional burnout will be reflected in self-perceived empathy at the end of the study.

Due to the novelty and curricular changes that its implementation would entail, the investigators want to quantify its effectiveness in the results sought, comparing the effectiveness of a face-to-face intervention, an online intervention with the same objectives and content, and a control group.

HYPOTHESIS:

1. Mean self-perceived empathy will increase at least 1 point in the face-to-face intervention group compared to the control group.
2. The professional burnout syndrome of the participants will be 10% lower in the face-to-face intervention group at the end of the study compared to the control group.
3. Personal skills (greater empathy, greater sense of coherence, greater resilience, internal locus of control, greater social support), will be independently inversely associated with the burnout syndrome, adjusting for personal factors (younger age, male sex, positive personality traits), organizational (less workload), training (greater adherence to the intervention, greater participation in other activities related to it) and by the participant's baseline anxiety and depression.
4. Face-to-face intervention will improve self-perceived empathy and decrease burnout syndrome better than online; these differences will be significant.

MAIN GOAL:

To evaluate the effectiveness of a face-to-face intervention in relation to its online counterpart and regular training according to changes registered in the degree of professional burnout syndrome and in self-rated empathy in residents of the Multiprofessional Teaching Units of Family Medicine and Community Nursing in Vigo, Zaragoza and Mallorca.

SECONDARY OBJECTIVES:

1. - Quantify the adjusted influence of the professional burnout syndrome on self-rated empathy.
2. - Quantify changes in resilience and their adjusted influence on the professional burnout syndrome.
3. - Quantify changes in the locus of control and their adjusted influence on the professional burnout syndrome.
4. - Quantify changes in social support and their adjusted influence on the professional burnout syndrome.
5. - Quantify changes in the sense of coherence and their adjusted influence on the professional burnout syndrome.

   MATERIAL AND METHODS

   Study design:

   Ante-post evaluation study of the effectiveness of an educational intervention to improve empathy, with three arms: face-to-face, online and control group, lasting 2 years. The intervention is organized during the training of residents of Family and Community Care in three teaching units in different health regions.

   Scope of study:

   In the face-to-face intervention group, 90 residents of the Vigo Family and Community Nursing Teaching Unit will participate, both Internal Resident Physicians (MIR) and Internal Resident Nurses (EIR), from the 2018, 2019, 2020 and 2021 promotions. In the online intervention, 70 (MIR and EIR) of Aragón Training Unit of the same promotions.

   In the control group, the same measurements were carried out on 180 residents, doctors and nurses, from the same classes of the Balearic Islands Teaching Unit, who agreed to participate in the study.

   Recruitment of participants:

   Residents will be informed of the existence of the study by people outside the research team. If they agree to be informed, they will be contacted and they will be explained what the study consists of, ensuring that their participation or rejection of it will not have any repercussions on their residence. Residents who agree to participate will accept the transfer of their contact details to the research team for their management by a specific professional of the Institute to which the resident belongs.

   The participants will be sent the surveys for completion on-line using the free software REDCap.

   Sample size:

   Under the hypothesis of achieving changes in the three components of the Copenhagen Burnout Inventory (CBI) similar to those achieved in the experience of the Harvard South Shore Psychiatry Residency Training Program (50), for alpha = 0.05 and beta = 0.80 and, With twice as many cases as controls, at least 74 residents are required in the intervention group and 148 in the control group (OpenEpi, version 3).

   Study period:

   The study will be conducted between November 2020 and June 2023.

   Randomization procedure (if applicable).

   Due to the characteristics of the intervention, it is not possible to randomize or use placebo. The registry will be masked and each participant will receive a random code that will not be known to any of the researchers. The masking and custody of the codes will be carried out by the data management unit of the Health Research Institute corresponding to the participant's area (Vigo, Zaragoza, Mallorca).

   Investigators conducting statistical analysis will be blind to group assignment.

   Measurements and interventions (main and secondary variables).

   Outcome variables: Self-rated empathy with Interpersonal Reactivity Index (IRI), level of burnout in the personal, work and relationship with clients spheres with the self-completed Copenhagen Burnout Inventory (CBI).

   Independent variables: Resilience measure with the abbreviated Connor-Davidson scale (10-item CD-RISC), self-perception of the Locus of control, perceived social support (Oslo-3) and the sense of coherence measured through the abbreviated Orientation to Life scale. Questionnaire (OLQ-13).

   Covariates: Sociodemographic (age, sex, nationality), profession, promotion, personality classification with TIPI-SP, baseline anxiety and depression measured through the Hospital Anxiety and Depression Scale (HADS) questionnaire, potentially stressful situations in the organization (average hours annual worked, average monthly shifts, number of patients / day in the primary care consultation), process indicators (number of workshops received, months of residence, months of stay in health center, hours of training in motivational interviewing and hours of training in mindfulness during residency and own iniciative).

   The completion of all the questionnaires takes an estimated time of 40 minutes and will be done at the beginning, the year and at the end of the project.

   The surveys will be carried out electronically. Participants will receive an e-mail with the link to access the online survey, which will be completed anonymously.

   In the first interface the participants will see the informed consent of the part of the survey, if they want to participate they will accept the terms and write their name, surname and reference teaching unit. These data will be transmitted independently of the survey results to the data management unit of the Health Research Institute of the participant's reference area. This will have a code that will be associated with the second interface, the questionnaire.

   In the second interface, the questionnaire will be displayed where they will have to answer the questions, with no answer being always possible.

   Description of the intervention

   Face-to-face intervention of the Vigo Teaching Unit:

   The intervention has been created specifically for this group, residents of Family and Community Medicine and Nursing, with the aim of acquiring or improving personal skills mediating in the processes of physical and mental well-being that help them face with more motivation, enthusiasm and personal resources professional challenges.

   It is based on conducting 4-hour face-to-face workshops every four months throughout the period of specialized health training. They will be instrumented through group dynamics, communication exercises, leadership, corporality, and reflective and emotional writing.

   Audiovisual media (videos, presentations, recordings) will be used. They will be developed face-to-face in a classroom equipped with the necessary means for training, including versatility of the space.

   The intervention has been developed by a family doctor, with training and experience in prevention and approach to individual factors that act as protective factors of "burnout". She herself will be the one who gives the workshops and is paid for it.

   The online intervention will pursue the same objectives and will be nourished by the same content as the face-to-face intervention. The theoretical contents will be adapted for online use, with the flexibility of access and organization that this entails for the participants, including videos, presentations, recordings ...

   Group techniques will be carried out online, every four months during the entire period of specialized health training. They will be instrumented through group dynamics, communication exercises, leadership, corporality, and reflective and emotional writing.

   The teacher and tutor responsible for the online intervention will be a member of the Aragonese team external to the teaching unit, a health psychologist with extensive training and experience in work and organizational psychology, as well as in clinical psychology.

   Control group:

   The control group will be made up of residents who start or have started their training in 2018, 2019, 2020 and 2021 of the Balearic Islands Teaching Unit.

   These residents will receive the usual training in communication skills, according to the program of their teaching unit. Once the study is completed, they will be able to enjoy the training with the best results, either in person or online.

   They will complete the same questionnaires at the beginning, at the year and at the end of the study, in the same periods as the intervention group and in the same agreed sequence.

   STATISTICAL METHODOLOGY

   The analyzes will be done by intention to treat, keeping all the participants in their initial group of membership, including the missing values through analysis of multiple imputations.

   The primary analysis will be the difference in means of empathy and the professional burnout syndrome, with multilevel generalized linear models. The dependent variables, the group, the baseline measurement of each dependent variable and the applicable covariates will be included; in addition, robust standard errors will be used.

   The following sensitivity analyzes will be carried out: 1) adjusting for the probability of the professional burnout syndrome at the baseline and those other covariates that could indicate an imbalance between the trial arms; 2) comparing unfit and tight models. Different definitions of compliance-adherence to interventions will also be used.

   All p values will be two-tailed and statistical significance will be considered at the ≤ 0.05 level. All intervals will be made at 95% confidence. For statistical analyzes, R.

   SAFETY AND ADVERSE EFFECTS:

   If through the responses to the questionnaires an imminent risk to the health of any of the participants is suspected, they will be informed of their results.

ELIGIBILITY:
Inclusion Criteria:

* Residents (doctors and nurses) of the three Family Medicine and Community Nursing Training Units
* From the 2018, 2019, 2020 and 2021 promotions
* Who want to participate in the study and signed informed consent.

Exclusion Criteria:

* Residents who refuse to participate and / or do not sign informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Self-rated empathy | Two years
  Interpersonal Reactivity Index, with four subscales, scores range from 0 to 28 in each one

SECONDARY OUTCOMES:
Self-rated burnout | Two years
  Copenhagen Burnout Inventory, with three subdimensions, ". Scores of 50 to 74 are considered 'moderate', 75-99 are high, and a score of 100 is considered severe burnout

CONTACTS AND LOCATIONS:
Overall Officials: Ana Clavería, MD, PhD, MPH, Principal Investigator — Sergas
Locations (1):
- Ana Clavería, Vigo, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 2023 to 2025
Access Criteria: Under request